CLINICAL TRIAL: NCT05062668
Title: Efficacy and Safety of iStent Inject and Inject W in the Management of Primary Open-angle Glaucoma
Acronym: EII
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: Central Hospital Saint Quentin (Other Government)
Responsible Party: Sponsor
Other Study IDs: PI2021_843_0191
Record Dates: First submitted 2021-09-21; First posted 2021-09-30 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: POAG; MIGS
Keywords: POAG; iStent inject; MIGS

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- iStent: POAG patient operated at the CHU of Amiens or the CH of Saint-Quentin of a combined cataract and iStent inject or inject W surgery from January 2018 to September 2020.
  Interventions: Procedure: cataract operation and istent
- cataract only: POAG patients operated only on cataract from January 2018 to September 2020.
  Interventions: Procedure: cataract operation only

INTERVENTIONS:
Procedure: cataract operation and istent — a cataract operation and the placement of one or two iStent inject or inject W at the same time
  Groups: iStent
Procedure: cataract operation only — Patients have a classic postoperative treatment after cataract.
  Groups: cataract only

SUMMARY:
Primary open-angle glaucoma (POAG) is a chronic eye disease in which the only validated treatment is to lower intraocular pressure (IOP). It is the 2nd leading cause of blindness worldwide. The iStent® inject and inject W is an implantable device that is part of a new entity of so-called minimally invasive glaucoma surgery whose goal is to lower IOP with minimal tissue disruption in order to avoid the complications of conventional glaucoma surgery. This surgery is used in conjunction with cataract surgery in France. The primary objective is to study the 1-year efficacy and safety of combined cataract and iStent inject and inject W in the management of POAG in an observational, retrospective, controlled study of a cohort of POAG patients undergoing cataract surgery only.

ELIGIBILITY:
Inclusion Criteria:

* patient who have undergone combined phacoemulsification surgery and insertion of at least one iStent® for chronic open-angle glaucoma in the ophthalmology department of the Amiens University Hospital or the Saint-Quentin University Hospital (iStent® group).
* patient who have undergone simple phacoemulsification surgery in a patient with chronic open-angle glaucoma in the ophthalmology department of the Amiens University Hospital (control group).
* patient with Chronic open-angle glaucoma confirmed by gonioscopic examination, visual field, optical coherence tomography of the optic nerve, fundus examination, pachymetry and intraocular air pressure and/or applanation.

Exclusion Criteria:

* acute angle closure glaucoma,
* chronic angle closure glaucoma,
* uveitic glaucoma,
* traumatic glaucoma,
* exfoliative glaucoma.
* Previous filtering surgery on the operated eye.
* Intraoperative complication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: There are two groups, the first group is the iStent group. The investigators took all the POAG patients operated at the CHU of Amiens or the CH of Saint-Quentin of a combined cataract and iStent inject or inject W surgery from January 2018 to September 2020. The second group is the control group of POAG patients operated only on cataract during the same period.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-10-08 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
variation of IOP (in mmHg) between both groups | 1 year
  variation of IOP (in mmHg) between the istent and cataract operation group versus the cataract operation only group

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Nord, Amiens, France

IPD SHARING:
Plan to Share IPD: No